CLINICAL TRIAL: NCT02925858
Title: Pilot Study: The Effect of Intraoperative Ketamine on Analgesia Post-Cardiac Surgery and Prevention of Chronic Pain
Brief Title: Effect of Ketamine on Analgesia Post-Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Matthew Cameron, Assistant Professor, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16-289
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Pain, Postoperative
Keywords: Ketamine; Cardiac surgery; Pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intraoperative infusion of ketamine
  Interventions: Drug: Ketamine Hydrochloride
- Control (Placebo Comparator): Control group receiving a saline infusion
  Interventions: Drug: Normal Saline Flush, 0.9% Injectable Solution_#1

INTERVENTIONS:
Drug: Normal Saline Flush, 0.9% Injectable Solution_#1 — Normal saline infusion mimicking infusion rate of ketamine for a given weight
  Arms: Control
Drug: Ketamine Hydrochloride — Ketamine IV infusion (0.5mg/kg bolus prior to incision, 0.5mg/kg/hr until the end of surgery)
  Arms: Intervention

SUMMARY:
Randomized, controlled, double-blind pilot study evaluating the effect of an intraoperative infusion of intravenous Ketamine on the quantity of opioid consumed postoperatively in coronary artery bypass surgery patients receiving a median sternotomy.

DETAILED DESCRIPTION:
This is a randomized, controlled, double-blind pilot study to determine the effectiveness of intraoperative Ketamine administration on pain after coronary artery bypass surgery. Patients will be randomized to receive ketamine or saline prior to incision, with a continuous infusion throughout surgery. Opioid dose administered in the first 48 hours will then be documented as the primary outcome

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older coming for coronary artery bypass surgery with a left ventricular ejection fraction over 50% and able to consent prior to surgery

Exclusion Criteria:

* Minimally invasive cardiac surgery
* Preoperative opioid use
* Preoperative hepatic or renal dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Cameron, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Will provide all uncoded data
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Upon request, starting 6 months after publication
Access Criteria: For planned meta-analyses

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 42 | 38
Completed | 42 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ketamine: Bolus 0.5mg/kg, Infusion 0.5mg/kg/hr
- Placebo: Normal Saline 0.025cc/kg bolus, 0.025cc/kg/hr
- Total: Total of all reporting groups
Arm/Group | Ketamine | Placebo | Total
Number analyzed (Participants) | 42 | 38 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (9.6) | 67.1 (8.6) | 66.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 38 | 33 | 71
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 42 | 38 | 80
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (4.2) | 28.0 (4.0) | 28.5 (4.1)
Cardiopulmonary Bypass time (mins) [Mean (Standard Deviation); unit: mins] | 105.4 (33.7) | 108.2 (29.6) | 106.7 (31.5)
Cross Clamp Time (mins) [Mean (Standard Deviation); unit: minutes] | 83.6 (33.4) | 82.7 (25.6) | 83.6 (33.4)
Intraoperative Sufentanil per kg [Mean (Standard Deviation); unit: mcg/kg] | 2.17 (1.11) | 1.96 (0.86) | 2.07 (1.07)

OUTCOME MEASURES:

1. Primary Outcome: Quantity of Opioids Used in the First 48 Hours Postoperatively
Description: Opioids used, in Dilaudid equivalents
Time Frame: First 48 hours after arrival to the ICU
Measure: Mean (95% Confidence Interval); unit: mg of Dilaudid
Groups:
- Ketamine: Intraoperative infusion of ketamine
  Ketamine Hydrochloride: Ketamine IV infusion (0.5mg/kg bolus prior to incision, 0.5mg/kg/hr until the end of surgery)
- Placebo: Control group receiving a saline infusion
  Normal Saline Flush, 0.9% Injectable Solution_#1: Normal saline infusion mimicking infusion rate of ketamine for a given weight
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 42 | 38
mg of Dilaudid | 10.71 [9.41 to 12.02] | 11.14 [9.68 to 12.61]

2. Secondary Outcome: Quantity of Opioids Used
Description: Quantity in mg
Time Frame: 24 hours postoperatively
Measure: Mean (95% Confidence Interval); unit: mg of Dilaudid
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 42 | 38
mg of Dilaudid | 6.5 [5.75 to 7.24] | 6.7 [5.94 to 7.45]

3. Secondary Outcome: Pain Scores (Visual Analog Scale)
Description: Average Pain Score as reported by the patient on a numeric scale ranging from 0 (no pain) to a maximum of 10 points (worst pain imaginable)
Time Frame: Postoperative days 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 42 | 38
score on a scale | 2 [0 to 4.25] | 2 [0 to 5]

4. Secondary Outcome: Postoperative Nausea and Vomiting
Description: Whether or not the patient suffered from nausea and vomiting after surgery which required treatment
Time Frame: 48 hours after ICU arrival
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 42 | 38
Participants | 3 | 2

5. Secondary Outcome: Intensive Care Unit Length of Stay
Description: Number of days spent in the intensive care unit
Time Frame: 1 day - 2 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 42 | 38
days | 1 [0 to 3] | 2 [0 to 4]

6. Secondary Outcome: Hospital Length of Stay
Description: number of days spent in the hospital, starting from the day of surgery
Time Frame: 5 days - 2 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 42 | 38
days | 8 [3 to 13] | 7 [2 to 12]

7. Secondary Outcome: Time to Extubation
Description: Number of minutes from the time of ICU arrival to extubation
Time Frame: 4 hours - 2 weeks
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 42 | 38
minutes | 539 [397 to 682] | 494 [383 to 605]

8. Secondary Outcome: Delirium
Description: Delirium as assessed by a positive CAM-ICU score during the ICU stay
Time Frame: ICU stay
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 42 | 38
Participants | 11 | 7

9. Secondary Outcome: Time to Mobilization
Description: Time from ICU arrival until patient able to mobilize to chair, measured in hours
Time Frame: During hospital stay
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 42 | 36
hours | 32 [26 to 40] | 23 [20 to 27]

10. Secondary Outcome: Time to Ambulation
Description: Time from ICU arrival until patient able to ambulate, measured in hours
Time Frame: 1 week postoperatively
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 42 | 36
hours | 63 [54 to 76] | 56 [46 to 64]

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Description: No noted adverse events
Arm/Group | Ketamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/38
Other Adverse Events (participants affected / at risk) | 0/42 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/58/NCT02925858/Prot_SAP_000.pdf